CLINICAL TRIAL: NCT00592605
Title: Thyroid Disease Serum Repository
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 84287
Record Dates: First submitted 2007-12-27; First posted 2008-01-14 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Thyroid disease is more common among females and is increasing in incidence.

Otolaryngology faculty members and residents will perform head and neck examinations as part of the subject's routine care. If the participant is noted to have thyroid disease, they will be asked if they would like to participate in the research portion by having approximately 10cc's of blood drawn. Faculty and staff will complete a data collection sheet that will contain demographic and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Participants with benign or malignant thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-05; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
To gather demographic and cultural information on approximately 1000 men and women with thyroid disease between the years 2007 and 2012 at the University of Arkansas for Medical Sciences. | 2007-2012

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Stack, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States